CLINICAL TRIAL: NCT05026034
Title: Correlation of the Non-invasive Cardiopulmonary Management (CPM) Wearable Device With Measures of Congestion in Heart Failure
Acronym: CONGEST HF
Status: Completed | Type: Observational
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Other Study IDs: GN20CA003
Record Dates: First submitted 2021-08-23; First posted 2021-08-30 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Wearable Electronic Devices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be taken for future cardiac biomarker analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Training Cohort: Inpatients with HF requiring >24 hours IV diuretics
  Interventions: Device: non-invasive Cardiopulmonary Management (CPM) wearable device
- Cohort A: Patients undergoing serial, clinically indicated RHC. To investigate if measures derived by the CPM wearable device correlate with invasive measures of cardiopulmonary haemodynamics (PCWP).
  Interventions: Device: non-invasive Cardiopulmonary Management (CPM) wearable device
- Cohort B: Patients receiving haemodialysis. To investigate if changes in measures derived by the CPM wearable device correlate with B-lines on LUS and changes in B-lines before and after haemodialysis and with volume of fluid removed during haemodialysis
  Interventions: Device: non-invasive Cardiopulmonary Management (CPM) wearable device
- Cohort C: Patients receiving inpatient intravenous diuretic treatment for heart failure. To investigate if changes in measures derived by the CPM wearable device system correlate with B-lines on lung ultrasound and weight before and after treatment for HF.
  Interventions: Device: non-invasive Cardiopulmonary Management (CPM) wearable device

INTERVENTIONS:
Device: non-invasive Cardiopulmonary Management (CPM) wearable device — non-invasive Cardiopulmonary Management (CPM) wearable device with measures of congestion in heart failure

SUMMARY:
Fluid status and congestion can be determined by the CPM wearable device and correlates with invasive measures, non-invasive measures and biochemical markers of congestion and changes in congestion.

DETAILED DESCRIPTION:
HF is associated with frequent and lengthy hospitalisations. These hospitalisations are usually as a result of congestion. The signs of congestion that can be recognised by physicians or health care professionals such as lung crackles or worsening of peripheral oedema are often seen at a late stage before an intervention can be made to prevent overt decompensation and admission to hospital. Recognising changes in excess fluid status either before a patient becomes unwell or during decongestion treatment is highly desirable so that timely treatment can be started or so that treatment can be adjusted based on an individual's response to therapy. The ability to assess patients by applying a single, non-invasive device would potentially provide a useful tool for assessing a patient's congestion levels and allow patients with progressive deterioration to be identified earlier.

ELIGIBILITY:
Inclusion Criteria:

Written informed consent

* Male or female over18 years of age Cohort A
* Meet European Society of Cardiology 1 (ESC) criteria for diagnosis of HF
* Undergoing clinically-indicated RHC Cohort B
* Established on haemodialysis for >90 days
* Undergoing haemodialysis with target volume removal ≥1.5 litres fluid Cohort C
* Meet ESC criteria for diagnosis of HF including heart failure
* Requiring treatment with intravenous (IV) diuretics Training Cohort
* Meet ESC criteria for diagnosis of HF including heart failure
* Requiring treatment with intravenous (IV) diuretics

Exclusion Criteria:

* Unable to consent to inclusion in study due to cognitive impairment
* Allergies or skin sensitivities to silicone-based adhesive
* Skin breakdown or dermatological condition on the left chest or breast areas or chest wall deformity where the device is placed
* Pregnancy or breast-feeding
* Conditions that may confound congestion assessments
* COVID-19 infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Heart Failure
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2022-07-22 (Actual)

PRIMARY OUTCOMES:
Cohort A: determine the correlation between congestion measured by the CPM wearable device and pulmonary capillary wedge pressure | 3 months
  Cohort A: determine the correlation between congestion measured by the CPM wearable device and pulmonary capillary wedge pressure measured in mmHg
Cohort B: To determine the correlation between congestion and change in congestion measured by the CPM wearable device and lung ultrasound (LUS) | 4 hours
  Cohort B: To determine the correlation between congestion and change in congestion measured by the CPM wearable device and lung ultrasound (LUS) measured as change in number of B lines
Cohort B: To determine the correlation between congestion and change in congestion measured by the CPM wearable device and lung ultrasound (LUS) | 4 hours
  Cohort B: To determine the correlation between congestion and change in congestion measured by the CPM wearable device and volume of fluid removed by dialysis in mls
Cohort C: To determine the correlation between congestion and change in congestion measured by the CPM wearable device and clinical measures of congestion | 24 hours
  Cohort C: To determine the correlation between congestion and change in congestion measured by the CPM wearable device and change in weight (kg)
Cohort C: To determine the correlation between congestion and change in congestion measured by the CPM wearable device and lung ultrasound (LUS) | 24 hours
  Cohort C: To determine the correlation between congestion and change in congestion measured by the CPM wearable device and lung ultrasound (LUS) measured as change in number of B lines

SECONDARY OUTCOMES:
Cohort A: To determine the correlation between pulmonary function measured by the CPM wearable device and spirometry | 24 hours
  Cohort A: To determine the correlation between pulmonary function measured by the CPM wearable device and spirometry measured by tidal volumes (ml/kg)
Cohort B: To determine the correlation between pulmonary function measured by the CPM wearable device and spirometry | 24 hours
  Cohort B: To determine the correlation between pulmonary function measured by the CPM wearable device and spirometry measured by tidal volumes (ml/kg)
Cohort C: To determine the correlation between pulmonary function measured by the CPM wearable device and spirometry | 24 hours
  Cohort C: To determine the correlation between pulmonary function measured by the CPM wearable device and spirometry measured by tidal volumes (ml/kg)
Cohort A: To determine the correlation between congestion measured by the CPM wearable device and the Everest clinical congestions score | 3 months
  Cohort A: To determine the correlation between congestion measured by the CPM wearable device and the Everest clinical congestions score grading 0 to 3 (with 0 being absent or a trace)
Cohort B: To determine the correlation between congestion measured by the CPM wearable device and the Everest clinical congestions score | 4 hours
  Cohort B: To determine the correlation between congestion measured by the CPM wearable device and the Everest clinical congestions score grading 0 to 3 (with 0 being absent or a trace)
Cohort C: To determine the correlation between congestion measured by the CPM wearable device and the Everest clinical congestions score | 24 hours
  Cohort C: To determine the correlation between congestion measured by the CPM wearable device and the Everest clinical congestions score grading 0 to 3 (with 0 being absent or a trace)
Cohort A: To determine the correlation between congestion measured by the CPM wearable device and right heart catheter (RHC) measurements | 3 months
  Cohort A: To determine the correlation between congestion measured by the CPM wearable device and right heart catheter (RHC) measurements
Cohort A: To determine the correlation between congestion measured by the CPM wearable device and echocardiography | 3 months
  Cohort A: To determine the correlation between congestion measured by the CPM wearable device and left ventricular ejection fraction (LVEF) measured as a percentrage by echocardiography
Cohort B: To determine the correlation between congestion measured by the CPM wearable device and echocardiography | 4 hours
  Cohort B: To determine the correlation between congestion measured by the CPM wearable device and left ventricular ejection fraction (LVEF) measured as a percentrage by echocardiography
Cohort C: To determine the correlation between congestion measured by the CPM wearable device and echocardiography | 24 hours
  Cohort C: To determine the correlation between congestion measured by the CPM wearable device and left ventricular ejection fraction (LVEF) measured as a percentrage by echocardiography

OTHER OUTCOMES:
Cohort A: Correlation coefficient between congestion score measured by CPM wearable device and NTproBNP | 3 months
  Cohort A: Correlation coefficient between congestion score measured by CPM wearable device and NTproBNP measured in pg/ml
Cohort B: Correlation coefficient between congestion score measured by CPM wearable device and NTproBNP | 4 hours
  Cohort B: Correlation coefficient between congestion score measured by CPM wearable device and NTproBNP measured in pg/ml
Cohort C: Correlation coefficient between congestion score measured by CPM wearable device and NTproBNP | 24 hours
  Cohort C: Correlation coefficient between congestion score measured by CPM wearable device and NTproBNP measured in pg/ml
Cohort A: Correlation coefficient between congestion score measured by CPM wearable device and change in haematocrit (Hct) | 3 months
  Cohort A: Correlation coefficient between congestion score measured by CPM wearable device and change in haematocrit (Hct) measured in L/L
Cohort B: Correlation coefficient between congestion score measured by CPM wearable device and change in haematocrit (Hct) | 4 hours
  Cohort B: Correlation coefficient between congestion score measured by CPM wearable device and change in haematocrit (Hct) measured in L/L
Cohort C: Correlation coefficient between congestion score measured by CPM wearable device and Change in haematocrit (Hct) | 24 hours
  Cohort C: Correlation coefficient between congestion score measured by CPM wearable device and Change in haematocrit (Hct) measured in L/L
Cohort C: Correlation coefficient between congestion score measured by CPM wearable device and left ventricular strain | 3 months
  Cohort C: Correlation coefficient between congestion score measured by CPM wearable device and left ventricular strain measured in percentage by echocardiography
Cohort C: Correlation coefficient between congestion score measured by CPM wearable device and right ventricular strain | 4 hours
  Cohort C: Correlation coefficient between congestion score measured by CPM wearable device and right ventricular strain measured in percentage by echocardiography
Cohort C: Correlation coefficient between congestion score measured by CPM wearable device and left atrial strain | 24 hours
  Cohort C: Correlation coefficient between congestion score measured by CPM wearable device and left atrial strain measured in percentage by echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Pardeep Jhund, Principal Investigator — Glasgow University and NHS Greater Glasgow and Clyde
Locations (2):
- United Kingdom (2):
  - Golden Jubilee National Hospital, Glasgow
  - Queen Elizabeth University Hospital, Glasgow

IPD SHARING:
Plan to Share IPD: Undecided
To be determined on completion of recruitment in line with sponsor policy